CLINICAL TRIAL: NCT05273281
Title: Pain-relieving Methods After Laparoscopic Hemicolectomy, Effects of Transabdominal Plain Block and Quadratus Lumborum Block
Brief Title: Pain-relieving Methods After Laparoscopic Hemicolectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R21075M
Record Dates: First submitted 2022-02-25; First posted 2022-03-10 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Pain; Nerve Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TAQLA (Experimental): Transabdominal plain block -group. Ropivacaine Hydrochloride Inj 5mg/ml 20 ml perineurally per side.
  Interventions: Procedure: Transabdominal plane block
- TAQLB (Experimental): Quadratus lumborum block -group. Ropivacaine Hydrochloride Inj 5mg/ml 20 ml perineurally per side.
  Interventions: Procedure: Quadratus lumborum block
- TAQLC (No Intervention): Control group. Pain relief only with intravenous and peroral drugs.

INTERVENTIONS:
Procedure: Transabdominal plane block — Peripheral nerve block
  Arms: TAQLA
Procedure: Quadratus lumborum block — Peripheral nerve block
  Arms: TAQLB

SUMMARY:
Effects of Transabdominal Plain Block and Quadratus Lumborum Block After Laparoscopic Hemicolectomy. The pain relief, bowel function and discharge.

DETAILED DESCRIPTION:
This study is proposed to explore the effects of transabdominal plane block and quadratus lumborum block after laparoscopic hemicolectomy.

After laparoscopic hemicolectomy there is a need for good analgesia. When the analgesia is adequate the patients mobilisation, bowel function and discharge is faster. Earlier, epidural block has been used for the analgesia but now the hemicolectomy is laparoscopic procedure and there is no need for central block anymore. Still patients needs opioids after the operation. Because of the opioids side effects, there is a need to find better analgesia methods.

In this study investigators compare peripheral nerve blocks, transabdominal plane and quadratus lumborum, for analgesia after laparoscopic hemicolectomy. Also investigators are comparing these analgesia methods and traditional orally analgesics. Patients receive transabdominal or quadratus lumborum block after induction using ropivacaine 5 mg/ml 20 ml per side. The third group is a control group witch analgesia is taken care with traditional orally analgesics.

After surgery investigators follow postoperative pain, opiate consumption, bowel function, nausea and mobilisation.

Investigators coal is to find if the transabdominal plain block or quadratus lumborum block prefer traditional analgesia methods after laparoscopic hemicolectomy.

ELIGIBILITY:
Inclusion Criteria:

Adult elective hemicolectomy patients

Exclusion Criteria:

Age under 18 years Complicated diabetes mellitus Lack of finnish language skill and/or co-operation Chronic pain Use of drugs that significantly influences the metabolism of paracetamol or opiate Steroid medication in regular use Significant liver-, lung- or kidney disfunction

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
First need of opiate | 72 hours or until discharge, whichever came first
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Opiate consumption | 72 hours or until discharge, whichever came first
  Total opiate consumption after surgery
Post operative pain | postoperatively: at 4 hours, at 8 hours,at 12 hours, at 16 hours, at 20 hours, at 24 hours, at 32 hours, 40 hours, at 48 hours, at 56 hours, at 64 hours, at 72 hours, ones per day after discharge for seven days after operation
  Numeric rating scale NRS 0-10, verbally description after discharge
Bowel function | postoperatively: at 4 hours, at 8 hours,at 12 hours, at 16 hours, at 20 hours, at 24 hours, at 32 hours, 40 hours, at 48 hours, at 56 hours, at 64 hours, at 72 hours, ones per day after discharge for seven days after operation
  Verbally description: non/gas/function
Nausea | postoperatively: at 4 hours, at 8 hours,at 12 hours, at 16 hours, at 20 hours, at 24 hours, at 32 hours, 40 hours, at 48 hours, at 56 hours, at 64 hours, at 72 hours, ones per day after discharge for seven days after operation
  Verbally description: yes/no

OTHER OUTCOMES:
Finnish pain query | Baseline and 4 week after operation
  This query has first made by the finnish association for the study of pain. It has been modified for this research. It includes questions how pain infects on the daily life (sleeping, exercising, ability to work, concentration et cetera), how often the pain appears and how intense the pain is (scale 0-10). There is a picture of body where patients marks the pain points.
Beck´s depression inventory (BDI) | Baseline and 4 week after operation
The State-Trait Anxiety Inventory (STAI) | Baseline and 4 week after operation

CONTACTS AND LOCATIONS:
Overall Officials: Jenni Kanerva, Phd, Principal Investigator — Tampere University Hospital; Maija-Liisa Kalliomäki, PhD, Study Director — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No